CLINICAL TRIAL: NCT05483517
Title: Efficacy of High Energy Density Pulse Electromagnetic Field for Patients With Rotator Cuff Tendinopathy: A Double-blinded, Randomized Controlled Trail
Brief Title: High Energy Density Pulse Electromagnetic Field for Patients With Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Liang-Cheng Chen, Director, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A202205076
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Rotator Cuff Tendinosis
Keywords: rotator cuff tendinopathy; high energy density pulse electromagnetic field
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy and high-PEMF (Experimental): The patient receives physiotherapy under the physiotherapist's guidance and high-PEMF therapy for three weeks, following two sessions a week.
  Interventions: Device: High energy density pulse electromagnetic field; Behavioral: physiotherapy
- physiotherapy and sham high-PEMF (Sham Comparator): The patient receives physiotherapy under the physiotherapist's guidance and sham high-PEMF therapy for three weeks, following two sessions a week.
  Interventions: Device: sham High energy density pulse electromagnetic field; Behavioral: physiotherapy

INTERVENTIONS:
Device: High energy density pulse electromagnetic field — The treatment coil is placed over the shoulder region at the maximum pain point for 9 minutes. A normal energy of high-PEMF with a rate of 2 pulse per second is applied to the patient.
  Arms: physiotherapy and high-PEMF
Device: sham High energy density pulse electromagnetic field — The sham treatment coil is placed over the shoulder region at the maximum pain point for 9 minutes. The setting is the same as the experimental group(normal energy, a rate of 2 pulse per second) with the difference that the energy output doesn't export to the patient.
  Arms: physiotherapy and sham high-PEMF
Behavioral: physiotherapy — Physiotherapy includes shoulder range of motion (ROM), stretching and muscle strengthening exercises. Under the physiotherapist's guidance, the patient receives the training session about 30 minutes every time.

SUMMARY:
The aim of our study is to investigate the efficacy of high energy density pulse electromagnetic field for patients with rotator cuff tendinopathy

DETAILED DESCRIPTION:
Traditional pulse electromagnetic field (PEMF) devices have been approved by the U.S. Food and Drug Administration (FDA) to treat nonunion fractures and cleared to treat post-operative pain and edema, osteoarthritis, and plantar fasciitis. However, high level of evidence indicated that the lack of beneficial effects of PEMF on pain, function or range of motion in the treatment of shoulder pain.

High energy density pulse electromagnetic field(High-PEMF) which builds up a voltage up to 30 kilovolt (kV) with shorter impulse time(50us) and broad band-width(200kHz~300MHz) is very different from traditional PEMF. Magnetic field about 50~150 millitesla (mT) is created and it can penetrate the body up to 20 cm. The aim of our study is to investigate the efficacy of High-PEMF for patients with rotator cuff tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 20 to 75 years old
2. persistent shoulder pain for at least 3 months and pain VAS score >=5
3. positive result in any of the following physical examinations: Hawkins-Kennedy, Neer or Jobe tests
4. confirmed rotator cuff tendinopathy by ultrasonography or MRI

Exclusion Criteria:

1. complete or full-thickness tear of rotator cuff found by ultrasonography or MRI
2. previous shoulder surgery
3. previous history of severe trauma in shoulder
4. cervical radiculopathy related shoulder pain or referred pain
5. other shoulder diseases: adhesive capsulitis, calcifying tendinopathy, radiology-confirmed acromion type III, shoulder instability, degenerative osteoarthritis, labral tear
6. present with any of the following systemic diseases: active infection, sever and uncontrolled medical condition, cancer, immune-related or rheumatoid arthritis, hyperuricemia and gout
7. previous treatment with articular or subacromial steroid injections within the last 3 months
8. cognitive impairment with loss of ability to sign the agreement and receive rehabilitation
9. pregnancy or lactating women
10. has any of the following contraindications: Carriers of pacemakers, internal defibrillators,internal metal implants (locally dependent), Cochlea implants, metallic stents, insulin pumps

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liang cheng Chen, MD, MS, Principal Investigator — Department of Physical Medicine and Rehabilitation, Tri-Service General
Locations (1):
- Tri-service general hospital, Taipei, Neihu, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Started | 12 | 12
Completed | 11 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 62.73 (7.51) | 56.10 (10.55) | 59.57 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 6 | 4 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 11 | 10 | 21
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 23.49 (2.11) | 23.47 (2.01) | 23.48 (2.01)
Duration (weeks) [Mean (Standard Deviation); unit: weeks] — The duration of shoulder pain before treatment.
  weeks | 13.91 (3.70) | 19.80 (14.91) | 16.71 (10.77)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Visual Analogue Scale(VAS)
Description: The Visual Analog Scale (VAS) was used to measure pain intensity. The scale ranges from 0 to 10, where 0 indicates no pain and 10 represents the worst possible pain. Higher scores indicate worse outcomes.
Time Frame: baseline, immediate after treatment, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Number analyzed (Participants) | 11 | 10
score on a scale
  baseline | 5.91 (2.51) | 5.90 (1.91)
  immediate after treatment | 4.73 (2.37) | 4.60 (2.27)
  4 weeks | 3.55 (1.69) | 4.90 (1.52)
  12 weeks | 3.72 (2.61) | 3.50 (1.27)

2. Secondary Outcome: Change in Total Score of Shoulder Pain and Disability Index (SPADI)
Description: The Shoulder Pain and Disability Index (SPADI) is a patient completed questionnaire with 13 items assessing pain level and extent of difficulty with activity of daily livings (ADLs) requiring the use of the upper extremities. The pain subscale has 5-items and the Disability subscale has 8-items. The patient is instructed to choose the number that best describes their level of pain and extent of difficulty using the involved shoulder. The pain scale is summed up to a total of 50 while the disability scale sums up to 80.
  The total SPADI score is calculated by adding the scores of the Pain and Disability subscales, with a range from 0 to 130. A higher total score indicates greater pain and disability.
Time Frame: baseline, immediate after treatment, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Number analyzed (Participants) | 11 | 10
score on a scale
  baseline | 58.27 (22.85) | 65.80 (32.25)
  immediate after treatment | 39.18 (25.13) | 52.40 (26.83)
  4 weeks | 41.27 (30.21) | 60.20 (41.16)
  12 weeks | 33.27 (21.28) | 30.80 (33.27)

3. Secondary Outcome: Changes of Shoulder Range of Motion in Active Flexion
Description: Shoulder ROM during flexion, abduction in the sitting position, internal rotation (IR) at 90° of abduction of the affected shoulder were measured using a digital goniometer, and the mean of three values was used for analysis
Time Frame: baseline, immediate after treatment, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Number analyzed (Participants) | 11 | 10
degree
  baseline | 143.74 (20.18) | 154.11 (23.47)
  immediately | 147.76 (19.81) | 152.53 (24.93)
  4 weeks | 144.89 (21.66) | 149.79 (24.70)
  12 weeks | 148.25 (22.54) | 159.29 (25.29)

4. Secondary Outcome: Changes of Shoulder Range of Motion in Active Abduction
Description: as for outcome 3
Time Frame: baseline, immediately after treatment, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Number analyzed (Participants) | 11 | 10
degree
  baseline | 142.51 (24.13) | 153.79 (26.34)
  immediately | 147.16 (24.78) | 154.22 (29.54)
  4 weeks | 152.93 (27.24) | 153.00 (28.30)
  12 weeks | 149.74 (25.48) | 163.34 (27.59)

5. Secondary Outcome: Changes of Shoulder Range of Motion in Active Internal Rotation
Description: as for outcome 3
Time Frame: baseline, immediately after treatment, 4 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
Number analyzed (Participants) | 11 | 10
degree
  baseline | 60.75 (18.71) | 73.03 (15.41)
  immediately | 68.46 (18.68) | 73.33 (14.33)
  4 weeks | 71.19 (15.56) | 80.94 (7.29)
  12 weeks | 76.66 (12.36) | 81.79 (11.29)

ADVERSE EVENTS:
Time Frame: 3 months
Description: no adverse event during treatment and follow up period
Arm/Group | Physiotherapy and High-PEMF | Physiotherapy and Sham High-PEMF
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05483517/Prot_SAP_000.pdf